CLINICAL TRIAL: NCT01444417
Title: A Phase 3 Randomized, Double Blind, Placebo Controlled Study to Determine the Safety and Efficacy of Romiplostim in Thrombocytopenic Pediatric Subjects With Immune Thrombocytopenia (ITP)
Brief Title: Safety and Efficacy Study of Romiplostim to Treat Immune Thrombocytopenia (ITP) in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20080279; 2010-018426-39 (EudraCT Number)
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Thrombocytopenia; Thrombocytopenia in Pediatric Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenia in Subjects With Immune (Idiopathic) Thrombocytopenic Purpura (ITP); Thrombocytopenic Purpura; Immune Thrombocytopenia
Keywords: Immune (Idiopathic) Thrombocytopenic Purpura; Pediatric Immune (Idiopathic) Thrombocytopenic Purpura; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura, Thrombocytopenic | interventions — romiplostim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Romiplostim (Experimental): Participants received once weekly subcutaneous romiplostim for 24 weeks at a starting dose of 1 µg/kg; weekly dose increases continued in increments of 1 µg/kg/week to a maximum dose of 10 µg/kg in an attempt to reach a target platelet count of ≥ 50 x 10^9/L.
  Interventions: Drug: Romiplostim
- Placebo (Placebo Comparator): Participants received weekly subcutaneous placebo for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Romiplostim — The starting dose of romiplostim is 1 µg/kg administered weekly by subcutaneous injection. Participants will return to the clinic weekly to provide platelet counts and undergo dose titrations under the supervision of the treating physician. Weekly dose increases will continue in increments of 1 µg/kg up to a maximum dose of 10 µg/kg in an attempt to reach a target platelet count of ≥ 50 x 10^9/L. Dose adjustment will be allowed during the treatment period to maintain a platelet count between ≥ 50 x 10^9/L and ≤ 200 x 10^9/L.
  Other Names: AMG 531; Nplate®
  Arms: Romiplostim
Drug: Placebo — Matching placebo administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of romiplostim in the treatment of thrombocytopenia in pediatric patients with Immune thrombocytopenia purpura (ITP) as measured by durable platelet response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary ITP according to the American Society of Hematology (ASH) guidelines at least 6 months prior to screening, regardless of splenectomy status
* Subject must be refractory to a prior ITP therapy, having relapsed after at least 1 prior ITP therapy, or ineligible for other ITP therapies; prior therapy includes first-line therapies
* Age ≥ 1 year and < 18 years at the time of providing informed consent
* The mean of 2 platelet counts taken during the screening period must be ≤ 30 x 10^9/L with neither count > 35 x 10^9/L
* A serum creatinine concentration ≤ 1.5 times the laboratory normal range (for each age category) during the screening period
* Adequate liver function; serum bilirubin ≤ 1.5 times the laboratory normal range during the screening period; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 times the laboratory normal range during the screening period
* Hemoglobin > 10.0 g/dL during the screening period
* Subject and/or subject's legally acceptable representative has provided informed consent prior to any study-specific procedure; subject has provided assent, where required

Exclusion Criteria:

* Known history of a bone marrow stem cell disorder; any abnormal bone marrow findings other than those typical of ITP must be approved by Amgen before a subject may be enrolled in the study
* Known active or prior malignancy except adequately treated basal cell carcinoma
* Known history of congenital thrombocytopenia
* Known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Known history of H. pylori by urea breath test or stool antigen test within 6 months of enrollment or successfully treated with no evidence of infection
* Known history of systemic lupus erythematosus, evans syndrome, or autoimmune neutropenia
* Known history of antiphospholipid antibody syndrome or positive for lupus anticoagulant
* Known history of disseminated intravascular coagulation, hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura
* Previous history of venous thromboembolism or thrombotic events
* Previous use of romiplostim, pegylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), Eltrombopag, recombinant human thrombopoietin (rHuTPO) or any platelet producing agent
* Rituximab (for any indication) or 6-mercaptopurine (6-MP) within 14 weeks before the screening visit, or anticipated use during the time of the proposed study
* Splenectomy within 4 weeks of the screening visit
* All hematopoietic growth factors including interleukin-11 (IL-11) (oprelvekin) within 4 weeks before the screening visit
* Alkylating agents within 8 weeks before the screening visit or anticipated use during the time of the proposed study
* Vaccinations known to decrease platelet counts within 8 weeks before the screening visit
* Known hypersensitivity to any recombinant E coli-derived product (eg, Infergen, Neupogen, Somatropin, and Actimmune)
* Other criteria may apply

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (24):
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, La Crosse, Wisconsin
- Australia (3):
  - Research Site, Randwick, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Parkville, Victoria
- Canada (4):
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec

REFERENCES:
- [Derived] Tarantino MD, Bussel JB, Blanchette VS, Despotovic J, Bennett C, Raj A, Williams B, Beam D, Morales J, Rose MJ, Carpenter N, Nie K, Eisen M. Romiplostim in children with immune thrombocytopenia: a phase 3, randomised, double-blind, placebo-controlled study. Lancet. 2016 Jul 2;388(10039):45-54. doi: 10.1016/S0140-6736(16)00279-8. Epub 2016 Apr 18. PMID 27103127
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 27 centers in the United States, Canada, and Australia. Participants were enrolled from 24 January 2012 to 03 September 2014.
Pre-assignment Details: Participants who met eligibility criteria were enrolled and stratified by the following 3 age categories: ≥ 1 to < 6 years; 6 to < 12 years; and 12 to < 18 years.
Period: Overall Study
Arm/Group | Placebo | Romiplostim
Started | 20 | 42
Received Treatment | 19 | 42
Completed | 18 | 41
Not Completed | 2 | 1
Not completed — Ineligibility Determined | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romiplostim | Total
Number analyzed (Participants) | 20 | 42 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (4.7) | 9.7 (4.1) | 9.6 (4.3)
Age, Customized [Number; unit: participants]
  ≥ 1 - < 6 years | 4 | 8 | 12
  ≥ 6 - < 12 years | 9 | 18 | 27
  ≥ 12 - < 18 years | 7 | 16 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 24 | 35
  Male | 9 | 18 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Black or African American | 2 | 6 | 8
  Multiple | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 1 | 5 | 6
  White | 15 | 26 | 41
Platelets [Mean (Standard Deviation); unit: 10^9/L] | 19.9 (19.3) | 17.5 (10.7) | 18.3 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Durable Platelet Response
Description: A participant with durable platelet response was defined as achieving at least 6 weekly platelet counts of ≥ 50 x 10^9/L during the last 8 weeks of treatment (platelet counts obtained from week 18 to week 25). If a platelet count from a participant was not available (missing) in a certain week, that week was imputed as non-response for that participant. Platelet counts were not deemed as a positive response for 4 weeks after the administration of rescue medication.
Time Frame: Week 18 to week 25
Population: Efficacy analysis set (all randomized participants)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 20 | 42
percentage of participants | 10.0 [1.2 to 31.7] | 52.4 [36.4 to 68.0]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; The incidence of durable platelet response was compared by the Cochran-Mantel-Haenszel test stratified by the baseline age group. The Mantel-Haenszel common odds ratio (romiplostim vs placebo) was estimated along with its 95% confidence interval; Test type: Superiority or Other; p = 0.0018, Cochran-Mantel-Haenszel; P-value from Cochran-Mantel-Haenszel test stratified by baseline age group; Odds Ratio (OR) = 9.0497, 95% CI 2-sided [1.896 to 43.199]

2. Secondary Outcome: Percentage of Participants With an Overall Platelet Response
Description: Overall platelet response is defined as either a durable platelet response or transient platelet response.
  Durable platelet response was defined as weekly platelet count ≥ 50 x 10^9/L for 6 or more times during week 18 to week 25 measurements. Participants may not have had a weekly response within 4 weeks after receiving any rescue medication.
  Transient platelet response was defined as weekly platelet count ≥ 50 x 10^9/L for 4 or more times during week 2 to week 25 measurements but without durable platelet response. Participants may not have had a weekly response within 4 weeks after receiving any rescue medications.
Time Frame: Week 2 to week 25
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 20 | 42
percentage of participants | 20.0 [5.7 to 43.7] | 71.4 [55.4 to 84.3]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; The incidence of overall platelet response was compared by the Cochran-Mantel-Haenszel test stratified by the baseline age group. The Mantel-Haenszel common odds ratio (romiplostim vs placebo) was estimated along with its 95% confidence interval; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; P-value from Cochran-Mantel-Haenszel test stratified by baseline age group; Odds Ratio (OR) = 9.0443, 95% CI 2-sided [2.535 to 32.265]

3. Secondary Outcome: Number of Weeks With Platelet Response
Description: Number of weeks with platelet counts ≥ 50 x 10^9/L during week 2 to week 25 measurements. Participants may not have had a weekly response within 4 weeks after receiving any rescue medications.
Time Frame: Week 2 to week 25
Population: Efficacy analysis set
Measure: Median (Full Range); unit: weeks
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 20 | 42
weeks | 1.0 [0 to 22] | 12.0 [0 to 24]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.0004, ANOVA; P-value from Analysis of Variance with main effects (treatment and age group) model after testing for non-significant interaction (p-value ≥ 0.10)

4. Secondary Outcome: Percentage of Participants Who Received Rescue Medication During the Treatment Period
Description: Rescue medication is any medication (other than excluded medications) that is intended to increase platelet counts or prevent bleeding.
Time Frame: 24 weeks
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 20 | 42
percentage of participants | 45.0 [23.1 to 68.5] | 40.5 [25.6 to 56.7]
Statistical Analysis 1: Comparison: Placebo vs Romiplostim; Test type: Superiority or Other; p = 0.7103, Cochran-Mantel-Haenszel; P-value from Cochran-Mantel-Haenszel test stratified by baseline age group; Odds Ratio (OR) = 0.813, 95% CI 2-sided [0.277 to 2.391]

5. Secondary Outcome: Total Number of Composite Bleeding Episodes
Description: A composite bleeding episode was defined as clinically significant bleeding events or the use of a rescue medication to prevent a clinical significant bleeding event during weeks 2 through 25 of the treatment period. A clinically significant bleeding event was defined as a Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 grade ≥ 2 bleeding event.
Time Frame: Week 2 to week 25
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: bleeding episodes
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 20 | 42
bleeding episodes | 4.0 (6.9) | 1.9 (4.2)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal,
  * life threatening (places the subject at immediate risk of death),
  * requires in-patient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity,
  * congenital anomaly/birth defect, and/or
  * other significant medical hazard. Adverse events were graded for severity according to the CTCAE version 3.0 grading scale, where Grade 3 = moderate, Grade 4 = life-threatening and Grade 5 = fatal.
  Treatment-related adverse events (TRAEs) were those assessed by the investigator as possibly related to study drug. This relationship was determined by a "yes" or "no" response to the question: "Is there a reasonable possibility that the event may have been caused by study drug?"
Time Frame: From the first dose of study drug until 4 weeks after last dose; 28 weeks.
Population: Safety analysis set (all participants who received at least one dose of study drug)
Measure: Number; unit: participants
Arm/Group | Placebo | Romiplostim
Number analyzed (Participants) | 19 | 42
participants
  Any adverse event (AE) | 19 | 41
  Serious adverse events (SAE) | 1 | 10
  AE leading to discontinuation of study drug | 0 | 0
  AE leading to discontinuation from study | 0 | 0
  Grade 3 AE | 3 | 6
  Grade 4 AE | 1 | 2
  Grade 5 AE | 0 | 0
  Treatment-related adverse events (TRAE) | 5 | 11
  Treatment-related serious adverse events | 0 | 1
  TRAE leading to discontinuation of study drug | 0 | 0
  TRAE leading to discontinuation from study | 0 | 0
  TRAE Grade 3 | 0 | 1
  TRAE Grade 4 | 0 | 0
  TRAE Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 4 weeks after last dose; 28 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romiplostim
Serious Adverse Events (participants affected / at risk) | 1/19 | 10/42
Other Adverse Events (participants affected / at risk) | 19/19 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Romiplostim (N=42)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Petit Mal Epilepsy (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Romiplostim (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Ear Pain (Ear and labyrinth disorders) | 2 | 2
Conjunctival Haemorrhage (Eye disorders) | 1 | 0
Scleral Discolouration (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival Bleeding (Gastrointestinal disorders) | 4 | 8
Lip Haemorrhage (Gastrointestinal disorders) | 1 | 2
Loose Tooth (Gastrointestinal disorders) | 1 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 4 | 11
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 8
Oral Disorder (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3
Tooth Socket Haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 4 | 11
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 7
Injection Site Bruising (General disorders) | 2 | 4
Injection Site Pain (General disorders) | 1 | 4
Localised Oedema (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 4
Peripheral Swelling (General disorders) | 0 | 4
Pyrexia (General disorders) | 2 | 9
Vessel Puncture Site Bruise (General disorders) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2
Oral Herpes (Infections and infestations) | 1 | 1
Pharyngitis Streptococcal (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 2 | 0
Sinusitis Bacterial (Infections and infestations) | 1 | 0
Tooth Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 16
Urinary Tract Infection (Infections and infestations) | 1 | 1
Viral Infection (Infections and infestations) | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Animal Scratch (Injury, poisoning and procedural complications) | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 21
Head Injury (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 6 | 2
Lip Injury (Injury, poisoning and procedural complications) | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Scratch (Injury, poisoning and procedural complications) | 2 | 6
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 4
Sunburn (Injury, poisoning and procedural complications) | 1 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Platelet Count Decreased (Investigations) | 3 | 5
Weight Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 11 | 17
Hypoaesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tension Headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depressed Mood (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Mood Altered (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 20
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 11
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Acne (Skin and subcutaneous tissue disorders) | 2 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 6
Rash Vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Mass (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 3
Tooth Extraction (Surgical and medical procedures) | 1 | 0
Haematoma (Vascular disorders) | 2 | 4
Haemorrhage (Vascular disorders) | 2 | 2
Pallor (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.